CLINICAL TRIAL: NCT00287001
Title: Effect of Cold Air Cooling on the Incidence of Post Inflammatory Hyperpigmentation Following a Q-Switched Nd:YAG Laser Treatment of Acquired Bilateral Nevus of Ota-Like Macules
Brief Title: Effect of Cold Air Cooling on the Incidence of Post Inflammatory Hyperpigmentation Following Laser Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Worapong Manuskiatti, Mahidol University
Allocation: Non-Randomized | Model: Single Group | Masking: Double
Other Study IDs: 185/2005
Record Dates: First submitted 2006-02-02; First posted 2006-02-06 (Estimated); Last update posted 2008-05-22 (Estimated); Status verified 2007-02

CONDITIONS: Nevus; Hyperpigmentation
Keywords: Acquired bilateral nevus of Ota-like macules; Postinflammatory hyperpigmentation; Cold air cooling
MeSH Terms: conditions — Nevus; Hyperpigmentation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Other): 1= cool air cooling
  Interventions: Device: Cold air cooling

INTERVENTIONS:
Device: Cold air cooling

SUMMARY:
- To investigate the benefit of epidermal cooling on the incidence of post inflammatory hyperpigmentation after laser irradiation

DETAILED DESCRIPTION:
* 70% incidence of post inflammatory hyperpigmentation has been reported following a Q-switched nd:YAG laser treatment of acquired bilateral nevus of Ota-like macules.
* We assumed that epidermal cooling may minimize the non-specific injury to the epidermis caused during laser irradiation, leading to the decreased incidence of post inflammatory hyperpigmentation.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with acquired bilateral nevus of Ota-like macules.
* At least 18 years old
* No previous treatment on the condition for a minimum period of 1 month.

Exclusion Criteria:

* Subjects diagnosed of scleroderma, connective tissue disorders, hematologic disorders, hepatitis, infection, or uncontrolled DM
* History of keloid and/or hypertrophic scar.
* Currently on anti-coagulant

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2005-12; Primary Completion 2006-04 (Actual); Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
Incidence of post inflammatory hyperpigmentation | 2 weeks

SECONDARY OUTCOMES:
Side effects of cold air cooling and clearing rate of pigmented lesion | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Woraphong - Manuskiatti, M.D., Principal Investigator — Mahidol University
Locations (1):
- Department of Dermatology, Siriraj Hospital, Mahidol University, Bangkok, Bangkok, Thailand

REFERENCES:
- [Background] Manuskiatti W, Sivayathorn A, Leelaudomlipi P, Fitzpatrick RE. Treatment of acquired bilateral nevus of Ota-like macules (Hori's nevus) using a combination of scanned carbon dioxide laser followed by Q-switched ruby laser. J Am Acad Dermatol. 2003 Apr;48(4):584-91. doi: 10.1067/mjd.2003.193. PMID 12664023
- [Background] Kunachak S, Leelaudomlipi P, Sirikulchayanonta V. Q-Switched ruby laser therapy of acquired bilateral nevus of Ota-like macules. Dermatol Surg. 1999 Dec;25(12):938-41. doi: 10.1046/j.1524-4725.1999.99176.x. PMID 10594626
- [Background] Raulin C, Grema H. Single-pass carbon dioxide laser skin resurfacing combined with cold-air cooling: efficacy and patient satisfaction of a prospective side-by-side study. Arch Dermatol. 2004 Nov;140(11):1333-6. doi: 10.1001/archderm.140.11.1333. PMID 15545541
- [Derived] Manuskiatti W, Eimpunth S, Wanitphakdeedecha R. Effect of cold air cooling on the incidence of postinflammatory hyperpigmentation after Q-switched Nd:YAG laser treatment of acquired bilateral nevus of Ota like macules. Arch Dermatol. 2007 Sep;143(9):1139-43. doi: 10.1001/archderm.143.9.1139. PMID 17875874